CLINICAL TRIAL: NCT03013842
Title: Feasibility of a Non-invasive, Trans-abdominal, Low Cost Fetal Oximetry Probe on Pregnant Human Subjects
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Principal Investigator no longer at Site
Sponsor: University of California, Davis (Other)
Collaborators: CITRIS (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 828902
Record Dates: First submitted 2016-12-05; First posted 2017-01-09 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Pregnancy, Abdominal
Keywords: pregnancy; fetal monitoring; fetal oximetry; fetal heart rate; pulse oximetry; near infrared spectroscopy
MeSH Terms: conditions — Pregnancy, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Administration of Fetal Oximetry Probe (Experimental): Administration of Raydiant Oximetry Sensor System on 36 weeks or greater pregnant women
  Interventions: Device: Raydiant Oximetry Sensor System

INTERVENTIONS:
Device: Raydiant Oximetry Sensor System — Administration of Fetal Oximetry Probe on 36 weeks or greater pregnant women
  Other Names: ROSS

SUMMARY:
Three non-invasive, trans-abdominal fetal oximetry probes will be tested on pregnant human subjects, in order to obtain fetal heart rate.

We want to determine if this device can accurately measure a baby's oxygen level when placed on your abdomen.

Current technology to measure a baby's oxygen levels requires a probe to be inserted into the vagina.

DETAILED DESCRIPTION:
The study subject will have a brief trans-abdominal ultrasound examination.

3 trans-abdominal fetal oximetry probes will be tested for 5 minutes per probe. No probes will be placed into the vagina.

It is anticipated that 6 months will be required to recruit, consent and study 25 participants.

ELIGIBILITY:
Inclusion Criteria:

* Greater than 36 weeks pregnant
* Singleton fetus

Exclusion Criteria:

* Prisoners

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2016-12-12 (Actual); Primary Completion 2017-08-02 (Actual); Study Completion 2017-08-02 (Actual)

PRIMARY OUTCOMES:
Fetal Photoplethysmogram | 6 months
  The primary outcome measure will be if a fetal photoplethysmogram is obtained in the time domain that correlates to the fetal heart rate.

SECONDARY OUTCOMES:
Fetal Heart Rate | 6 months
  The secondary endpoint will be if fetal heart rate can be obtained in the frequency domain that correlates to a fetal heart rate obtained by Doppler.

CONTACTS AND LOCATIONS:
Overall Officials: Neil Ray, MD, Principal Investigator — 916-734-5028
Locations (1):
- University of California, Davis Medical Center, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No